CLINICAL TRIAL: NCT06162338
Title: A Prospective, Single-center, Open-arm, Single-arm Study of the Safety and Preliminary Efficacy of Single Intravenous Infusion Administration of LY-M001 Injection in the Treatment of Adult Patients with Gaucher Disease Type I
Brief Title: A Study of the Safety and Preliminary Efficacy of LY-M001 Injection in the Treatment of Adult Patients with Gaucher Disease Type I
Acronym: LY-M001
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: He Huang (Other)
Collaborators: Lingyi Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, He Huang, Chief physician, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LY-M001-GD-001
Record Dates: First submitted 2023-11-20; First posted 2023-12-08 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Gaucher Disease Type I
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Intervention Model Description: A Prospective, Single-center, Open-label, Single-arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- A Prospective, single-center, open, single-arm study (Experimental): The study is single-arm. LY-M001 injection is administered by intravenous infusion at a rate of 1 mL per minute.LY-M001 Injection is Clear and colorless liquid.According to the dose cohort of the subject, the required dosage was accurately calculated by the patient's body weight for infusion.
  Interventions: Biological: LY-M001 Injection

INTERVENTIONS:
Biological: LY-M001 Injection — With 5.0 × 10^12 vg/kg as the initial effective dose (first dose group), 1 to 2 subjects are expected to be included. The first dose group was enrolled by sentinel method, and the first subject in this group was observed for at least 28 days after receiving LY-M001 (dose-limited toxicity [DLT] observation period) to enroll the next subject. After the first participant completes the safety evaluation of dosing for at least 28 days, the investigator (PI) and the partner discuss the safety and efficacy data and decide to maintain the first dose or increase/reduce it to another dose group

SUMMARY:
This is a prospective single-center, open, single-arm, single-dose intravenous infusion study to evaluate the safety and initial efficacy, pharmacodynamic characteristics, immunogenicity, biodistribution, and viral shedding of LY-M001 injection.This study mainly includes the main study stage and the long-term follow-up study stage.

DETAILED DESCRIPTION:
This study included the screening period (weeks -8 to days -2), the baseline period (days -1), the treatment and safety observation period (days 0 to 28), and the short-term follow-up period (weeks 5 [from day 29] to week 38). Participants eligible for the screening period will be admitted to the study center for a single LY-M001 treatment and a short-term follow-up period after the end of the treatment and safety observation period. Participants who complete all follow-up during the main study phase or who withdraw early from the study are required to complete all assessments required for the End of Study (EOS) visit.The study included up to three adult Gaucher disease type I subjects at preset dose group levels.With 5.0 × 1012 vg/kg as the initial effective dose (first dose group), 1 to 2 subjects are expected to be included. The first dose group was enrolled by sentinel method, and the first subject in this group was observed for at least 28 days after receiving LY-M001 (dose-limited toxicity [DLT] observation period) to enroll the next subject.

Participants enrolled in the long-term follow-up study were those who completed the main study or withdrew early, and the duration of the long-term follow-up study and the main study lasted for a total of 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤ 60 years, male or female.
2. The subjects should fully understand the purpose, nature and method of this study as well as possible adverse reactions, and sign the informed consent form (ICF) voluntarily.
3. Patients with GD1 who have confirmed double mutations in the Gba1 allele by laboratory testing and meet the standard for clinical diagnosis of Gaucher disease (i.e., reduced GCase enzyme activity to less than 30% of normal values).
4. The subjects were type I patients with Gaucher disease. Patients with type I Gaucher disease who had received specific treatment in the past required 5 half-lives of elution
5. Negative pregnancy test for female subjects of childbearing potential 6.6.The subject and his/her partner have no plans to have children during the screening period and within 6 months after the end of the study, and voluntarily take effective contraceptive measures (such as abstinence, condom, etc.); and the subject had no plans to donate sperm or eggs.

7.Subjects are not to donate blood during the study and for at least 1 year after the end of the study.

Exclusion Criteria:

1. AAV8 neutralizing antibody is strongly positive.
2. Patients with clinically suspected Gaucher disease type II (GD2) or Gaucher disease type III (GD3).
3. Active and progressive bone disease that is expected to require surgical treatment within the next 6 months.
4. Subject has idiopathic thrombocytopenic purpura (ITP), thrombotic thrombocytopenic purpura (TTP), thrombocytopenia, anemia, hepatomegaly, splenomegaly, and/or osteoporosis unrelated to Gaucher disease as judged by the investigator.
5. Treatment or disposition of an investigational drug or investigational device for another clinical investigation within 28 days or 5 half-lives (only for drugs), whichever is longer, prior to Screening.
6. Evidence of clinically significant liver disease, fragile liver, or history of hepatotoxin exposure, meeting at screening, but not limited to, any of the following:

   * Progressive hepatomegaly and greater than 3 times normal volume.
   * History of stage 2 or greater liver fibrosis.
   * AST, ALT or TBIL greater than 1.5 times the upper limit of normal (ULN).
   * History of alcohol or drug abuse within the previous 2 years.
   * Hepatitis B surface antigen (HBsAg) positive, and hepatitis B virus DNA positive (HBV-DNA > 103 copies/mL); or taking hepatitis B virus drugs (such as interferon, lamivudine, adefovir and entecavir); or hepatitis C virus (HCV) antibody positive.
7. Human immunodeficiency virus (HIV) antibody positive or Treponema pallidum antibody positive.
8. Severe hyperlipidemia (triglycerides > 1000 mg/dL).
9. Uncontrolled concomitant disease or infectious disease (need to be judged by the investigator based on clinical practice).
10. Subject had undergone splenectomy and were scheduled to undergo splenectomy during the study period.
11. Karnofsky score (KPS) < 70.
12. The subject has received or plans to receive bone marrow transplantation, hematopoietic stem cell transplantation and/or major organ transplantation, including but not limited to liver transplantation, kidney transplantation, etc.
13. Subject has received erythropoietin, transfusion, or red blood cell transfusion within 3 months prior to screening ;or platelet transfusion within 1 month prior to screening.
14. Clinically diagnosed or significant cardiovascular disease as judged by the investigator (e.g., New York Heart Association [NYHA] class ≥ 3 heart failure).
15. Hypersensitivity to any component of LY-M001 Injection.
16. Previous treatment with any type of gene therapy or cell therapy.
17. Use of systemic immunosuppressive agents or steroid therapy other than those required by the protocol for prophylactic administration within 3 months prior to dosing.
18. History of cancer within 5 years of screening, except for completely resected non-melanoma skin cancer, non-metastatic prostate cancer, and completely treated ductal carcinoma in situ.
19. Has received a live attenuated vaccine within 4 months prior to screening or plans to receive a live attenuated vaccine during the clinical trial.
20. Other conditions that, in the opinion of the investigator, make the subject unsuitable for the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2026-12-17 (Estimated); Study Completion 2031-12-17 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment- related adverse events | within 38 weeks after LY-M001 infusion
  Number and severity of adverse events and serious adverse events and relationship to LY-M001
Incidence of events adjudicated as dose limiting toxicity (DLT) | within 28 days after LY-M001 infusion
  Number and severity of dose limiting toxicity

SECONDARY OUTCOMES:
Glucocerebrosidase (GCase) protein in plasma and GCase enzyme activity | Within 38 Weeks after LY-M001 infusion
  Change from baseline in plasma GCase protein and GCase enzyme activity level
Glucosylsphingosine (Lyso-GL1)in plasma | Within 38 Weeks after LY-M001 infusion
  Change from baseline in plasma Lyso-GL1 level

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang University School of Medicine, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nabizadeh A, Amani B, Kadivar M, Toroski M, Asl AA, Bayazidi Y, Mojahedian M, Davari M. The Clinical Efficacy of Imiglucerase versus Eliglustat in Patients with Gaucher's Disease Type 1: A Systematic Review. J Res Pharm Pract. 2018 Oct-Dec;7(4):171-177. doi: 10.4103/jrpp.JRPP_18_24. PMID 30622983
- [Background] Barranger JA, Brady RO, Grabowski GA, Mankin H, Mistry PK, Weinreb NJ. Position statement: National Gaucher Foundation Medical Advisory Board, January 7, 2014. Am J Hematol. 2014 May;89(5):457-8. doi: 10.1002/ajh.23687. Epub 2014 Mar 7. No abstract available. PMID 24488939
- [Background] Franco M, Reihani N, Marin M, De Person M, Billette de Villemeur T, Rose C, Colin Y, Moussa F, Belmatoug N, Le Van Kim C. Effect of velaglucerase alfa enzyme replacement therapy on red blood cell properties in Gaucher disease. Am J Hematol. 2017 Sep;92(9):E561-E563. doi: 10.1002/ajh.24816. Epub 2017 Jul 19. No abstract available. PMID 28621801
- [Background] Kuter DJ, Wajnrajch M, Hernandez B, Wang R, Chertkoff R, Zimran A. Open-label, expanded access study of taliglucerase alfa in patients with Gaucher disease requiring enzyme replacement therapy. Blood Cells Mol Dis. 2020 May;82:102418. doi: 10.1016/j.bcmd.2020.102418. Epub 2020 Feb 24. PMID 32146279
- [Background] Bennett LL, Fellner C. Pharmacotherapy of Gaucher Disease: Current and Future Options. P T. 2018 May;43(5):274-309. PMID 29719368
- [Background] Tsai P, Lipton JM, Sahdev I, Najfeld V, Rankin LR, Slyper AH, Ludman M, Grabowski GA. Allogenic bone marrow transplantation in severe Gaucher disease. Pediatr Res. 1992 May;31(5):503-7. doi: 10.1203/00006450-199205000-00019. PMID 1603628
- [Background] Konkle BA, Walsh CE, Escobar MA, Josephson NC, Young G, von Drygalski A, McPhee SWJ, Samulski RJ, Bilic I, de la Rosa M, Reipert BM, Rottensteiner H, Scheiflinger F, Chapin JC, Ewenstein B, Monahan PE. BAX 335 hemophilia B gene therapy clinical trial results: potential impact of CpG sequences on gene expression. Blood. 2021 Feb 11;137(6):763-774. doi: 10.1182/blood.2019004625. PMID 33067633
- [Background] Nathwani AC, Reiss UM, Tuddenham EG, Rosales C, Chowdary P, McIntosh J, Della Peruta M, Lheriteau E, Patel N, Raj D, Riddell A, Pie J, Rangarajan S, Bevan D, Recht M, Shen YM, Halka KG, Basner-Tschakarjan E, Mingozzi F, High KA, Allay J, Kay MA, Ng CY, Zhou J, Cancio M, Morton CL, Gray JT, Srivastava D, Nienhuis AW, Davidoff AM. Long-term safety and efficacy of factor IX gene therapy in hemophilia B. N Engl J Med. 2014 Nov 20;371(21):1994-2004. doi: 10.1056/NEJMoa1407309. PMID 25409372
- [Background] Xu YH, Quinn B, Witte D, Grabowski GA. Viable mouse models of acid beta-glucosidase deficiency: the defect in Gaucher disease. Am J Pathol. 2003 Nov;163(5):2093-101. doi: 10.1016/s0002-9440(10)63566-3. PMID 14578207
- [Background] Sun Y, Zhang W, Xu YH, Quinn B, Dasgupta N, Liou B, Setchell KD, Grabowski GA. Substrate compositional variation with tissue/region and Gba1 mutations in mouse models--implications for Gaucher disease. PLoS One. 2013;8(3):e57560. doi: 10.1371/journal.pone.0057560. Epub 2013 Mar 8. PMID 23520473
- [Background] Chen RL, Hou JW, Chang PY, Tsai FJ, Wang PJ. Matched unrelated bone marrow transplantation without splenectomy for a child with Gaucher disease caused by homozygosity of the L444P mutation, who also suffered from schizencephaly. J Pediatr Hematol Oncol. 2007 Jan;29(1):57-9. doi: 10.1097/MPH.0b013e3180308793. PMID 17230068
- [Background] Chowdary P, Shapiro S, Makris M, Evans G, Boyce S, Talks K, Dolan G, Reiss U, Phillips M, Riddell A, Peralta MR, Quaye M, Patch DW, Tuddenham E, Dane A, Watissee M, Long A, Nathwani A. Phase 1-2 Trial of AAVS3 Gene Therapy in Patients with Hemophilia B. N Engl J Med. 2022 Jul 21;387(3):237-247. doi: 10.1056/NEJMoa2119913. PMID 35857660
- See also: A Phase I/II, Open label, Multicentre, Ascending Single Dose, Safety Study of a Novel Adeno associated Viral Vector (FLT180a) in Patients With Haemophilia B 2020 — http://clinicaltrials.gov/ProvidedDocs/44/NCT03369444/Prot_001.pdf
- See also: Package Insert - HEMGENIX — http://www.fda.gov/vaccines-blood-biologics/vaccines/hemgenix
- See also: WHOQOL - Files — http://iris.who.int/bitstream/handle/10665/77932/WHO_HIS_HSI_Rev.2012.03_eng.pdf